CLINICAL TRIAL: NCT01833936
Title: The Use of Electrical Stimulation on Muscle Cross Sectional Area and Muscle Fascicle Length Following Postoperative Achilles Tendon Repair
Brief Title: E-Stim and Achilles Tendon Repair Study
Acronym: E-Stim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedic Foot and Ankle Center, Ohio (Other)
Collaborators: DonJoy Orthotics (Industry)
Responsible Party: Principal Investigator, Christopher Hyer, DPM, MS, Orthopedic Foot and Ankle Center, Ohio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OH1-12-00389
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1- Compex® muscle stimulator (Active Comparator): Group 1 will receive an active muscle stimulator, which will be placed immediately following surgery. Eight electrodes will be placed on the lower leg: four electrodes on the gastrocnemius (calf muscle), and two electrodes each on the lateral gastrocnemius (side) and anterior tibialis muscle (front). Subjects will use the stimulator for three 20 minute sessions per day.
  Interventions: Device: Compex® muscle stimulator
- Group 2 -(inactive) muscle stimulator (Sham Comparator): Group 2 will receive a placebo (inactive) muscle stimulator, which will be placed immediately following surgery. Eight electrodes will be placed on the lower leg: four electrodes on the gastrocnemius (calf muscle), and two electrodes each on the lateral gastrocnemius (side) and anterior tibialis muscle (front). Subjects will be instructed to use the stimulator for three 20 minute sessions per day.
  Interventions: Device: (inactive) muscle stimulator

INTERVENTIONS:
Device: Compex® muscle stimulator — The Compex® muscle stimulator is a commercially available muscle stimulator that is approved by the Food and Drug Administration (FDA), a governmental body. It is not investigational. The investigational part of this study aims to evaluate if the use of muscle simulation after Achilles tendon surgery will reduce calf atrophy.
  Arms: Group 1- Compex® muscle stimulator
Device: (inactive) muscle stimulator — A placebo (inactive) muscle stimulator, which will be placed immediately following surgery. Eight electrodes will be placed on the lower leg: four electrodes on the gastrocnemius (calf muscle), and two electrodes each on the lateral gastrocnemius (side) and anterior tibialis muscle (front). Subjects will be instructed to use the stimulator for three 20 minute sessions per day.
  Arms: Group 2 -(inactive) muscle stimulator

SUMMARY:
Calf muscle atrophy (muscle degeneration) is common following Achilles tendon repair due to the immobilization period necessary to ensure optimal healing.

The purpose of this study is to determine if the use of neuromuscular electrical stimulation (NMES) after Achilles tendon surgery will reduce calf muscle atrophy.

DETAILED DESCRIPTION:
The specific aims of this study are to evaluate the use of electrical stimulation on muscle cross-sectional area and muscle fascicle length following post-operative Achilles tendon surgery.

Patients will be randomly assigned to receive an electrical stimulation unit (Compex®, DJO Global, San Diego, CA). Twenty of these units will be experimental and 20 will be sham.

ELIGIBILITY:
Inclusion Criteria:

* 1. Any patient who is having surgery to treat an acute Achilles tendon rupture or any surgery that involves reflecting or repairing the distal Achilles tendon.

Exclusion Criteria:

1. Body mass index (BMI) greater than or equal to 45
2. Inability to consent to participate in clinical research
3. Any patient younger than 18 years old
4. Any limitations that would interfere with the delivery of electrical stimulation including, but not limited to:

   1. Presence of an insulin pump
   2. Pacemaker, defibrillators or other implanted electrical device
   3. Neurostimulation implants
   4. History of epilepsy/seizure
   5. Current pregnancy. A pregnancy test will be performed for any female prior to surgical intervention per hospital protocol unless she is post-menopausal or has been sterilized.
   6. Active malignancy
   7. Peripheral neuropathy
   8. Diabetes Mellitus
   9. Ischemia of lower limbs
   10. Active infection
   11. Following acute trauma or fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2016-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hyer, DPM, MS, Principal Investigator — Orthopedic Foot and Ankle Center
Locations (1):
- Orthopedic Foot and Ankle Center, Westerville, Ohio, United States

REFERENCES:
- [Background] Gomes AR, Cornachione A, Salvini TF, Mattiello-Sverzut AC. Morphological effects of two protocols of passive stretch over the immobilized rat soleus muscle. J Anat. 2007 Mar;210(3):328-35. doi: 10.1111/j.1469-7580.2007.00697.x. PMID 17331181
- [Background] Gorodetskyi IG, Gorodnichenko AI, Tursin PS, Reshetnyak VK, Uskov ON. Use of noninvasive interactive neurostimulation to improve short-term recovery in patients with surgically repaired bimalleolar ankle fractures: a prospective, randomized clinical trial. J Foot Ankle Surg. 2010 Sep-Oct;49(5):432-7. doi: 10.1053/j.jfas.2010.05.007. Epub 2010 Aug 5. PMID 20688546
- [Background] Lieber RL, Ward SR. Skeletal muscle design to meet functional demands. Philos Trans R Soc Lond B Biol Sci. 2011 May 27;366(1570):1466-76. doi: 10.1098/rstb.2010.0316. PMID 21502118
- [Background] Takano Y, Haneda Y, Maeda T, Sakai Y, Matsuse H, Kawaguchi T, Tagawa Y, Shiba N. Increasing muscle strength and mass of thigh in elderly people with the hybrid-training method of electrical stimulation and volitional contraction. Tohoku J Exp Med. 2010 May;221(1):77-85. doi: 10.1620/tjem.221.77. PMID 20453461

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1- Compex® Muscle Stimulator | Group 2 -(Inactive) Muscle Stimulator
Started | 20 | 20
Completed | 16 | 18
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1- Compex® Muscle Stimulator | Group 2 -(Inactive) Muscle Stimulator | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (9.6) | 45.8 (11.8) | 48.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.4 (5.6) | 31.1 (5.6) | 32.2 (5.7)
Tobacco Use [Count of Participants; unit: Participants]
  Current | 2 | 1 | 3
  Former | 4 | 2 | 6
  Never | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Reduce Calf Muscle Atrophy
Description: Magnetic resonance imaging (MRI) scans were conducted preoperatively and postoperatively at weeks 2 and 6 to measure cross sectional muscle volumes of the calf muscle. By measuring the muscle volume, the investigators hope to show the use of electrical stimulation will reduce calf muscle atrophy.
Time Frame: Pre-operative, 2 weeks, and 6 weeks post-operative
Population: Pre-operatively, 20 subjects were analyzed per arm. Due to subject withdrawal, 19 were available in Group 1 at 2 weeks; and only 16 were available in Group 1 at 6 weeks, and 10 were available in Group 2 at 6 weeks.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Group 1- Compex® Muscle Stimulator | Group 2 -(Inactive) Muscle Stimulator
Number analyzed (Participants) | 20 | 20
mm^2
  Pre-operative Lateral Gastrocnemius | 859.8 (230.1) | 874.9 (228.4)
  Pre-operative Medial Gastrocnemius | 1450.4 (392.1) | 1634.9 (378.2)
  Pre-operative Soleus | 1962.2 (456.6) | 2250.5 (701.9)
  2 weeks post-operative Lateral Gastrocnemius: number analyzed (Participants) | 19 | 20
  2 weeks post-operative Lateral Gastrocnemius | 754.5 (184.4) | 780.9 (217.3)
  2 weeks post-operative Medial Gastrocnemius: number analyzed (Participants) | 19 | 20
  2 weeks post-operative Medial Gastrocnemius | 1348.1 (420.7) | 1432.8 (324.0)
  2 weeks post-operative Soleus: number analyzed (Participants) | 19 | 20
  2 weeks post-operative Soleus | 1835.7 (461.0) | 2057.0 (646.7)
  6 weeks post-operative Lateral Gastrocnemius: number analyzed (Participants) | 16 | 10
  6 weeks post-operative Lateral Gastrocnemius | 729.4 (195.6) | 722.9 (191.6)
  6 weeks post-operative Medial Gastrocnemius: number analyzed (Participants) | 16 | 10
  6 weeks post-operative Medial Gastrocnemius | 1242.1 (418.6) | 1316.2 (309.7)
  6 weeks post-operative Soleus: number analyzed (Participants) | 16 | 10
  6 weeks post-operative Soleus | 1780.3 (471.3) | 1907.5 (586.4)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Group 1- Compex® Muscle Stimulator | Group 2 -(Inactive) Muscle Stimulator
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/20
Other Adverse Events (participants affected / at risk) | 9/20 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- Compex® Muscle Stimulator (N=20) | Group 2 -(Inactive) Muscle Stimulator (N=20)
Achilles Tendon Re-ruptured (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject fell and re-ruptured Achilles tendon, which required additional surgery
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Subject was positive for deep vein thrombosis.
MRSA infection (Infections and infestations) | 0 (0) | 1 (1) — Subject had surgery on 08/10/2016. Subject return to clinic with increased pain, redness, and swelling. Subject went to ER also. Cultures positive for MRSA.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- Compex® Muscle Stimulator (N=20) | Group 2 -(Inactive) Muscle Stimulator (N=20)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
Achilles Incision irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Severe muscle discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject stated "felt like jumping out of my skin".
Achilles wound dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Increased ankle pain due to fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Skin irritation around electrode pads (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Knee pain and clicking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tooth pain (General disorders) | 0 (0) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Non-infected clear discharge from Achilles incision (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diagnosed with Bell's Palsy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No